CLINICAL TRIAL: NCT05889572
Title: Safety, Tolerability and Gut microbIota AnalysiS of an Oral Microbiotherapy in Amyotrophic Lateral Sclerosis; an Open-label Phase 1b Pilot Trial
Brief Title: Safety and Gut Microbiota Analysis of an Oral Microbiotherapy in Patients With Amyotrophic Lateral Sclerosis
Acronym: IASO
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: MaaT Pharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MPNS01
Record Dates: First submitted 2023-04-17; First posted 2023-06-05 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Amyotrophic Lateral Sclerosis; ALS
Keywords: Microbiotherapy; Amyotrophic Lateral Sclerosis; Neurodegenerative disease; ALS
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis; Neurodegenerative Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- MaaT033 (Experimental): Route of administration: oral (capsule)
  Between D-5 to D-1: Bowel preparation with Macrogol and Rifamixin
  Between D1 to D28: MaaT033 treatment period 1
  Between D28 to D56: MaaT033 treatment period 2
  Interventions: Drug: MaaT033

INTERVENTIONS:
Drug: MaaT033 — MaaT033 is a Microbiome Ecosystem Therapy (MET), composed of allogeneic, full-ecosystem pooled biotherapeutic gut microbiota.

SUMMARY:
The purpose of this pilot study is to assess the safety and tolerability of multiple doses of MaaT033 in ALS patients and to analyze the gut microbiota composition and evolution before considering a larger randomized controlled efficacy study.

DETAILED DESCRIPTION:
This is a prospective, single arm, open-label study.

The target population includes subjects with a recent disease onset defined as the time from first motor deficit at screening of at least 6 months and up to 24 months and removing very rapid/slow progressors based on the ALS Functional Rating Scale - Revised (ALSFRS-R) progression slope.

After a screening period (clinical examination, blood sampling), subject will come for a baseline visit (clinical examination, blood and feces sampling) and to initiate a bowel preparation phase. Five days later, subject will come back to the study site (clinical examination, blood sampling) to initiate a first Maat033 treatment period of 28-day. Ten days after MaaT033 treatment initiation a remote visit is included (feces sampling) to check the subject safety/tolerability. After the first Maat033 treatment period, subject will come to the study site (clinical examination, blood and feces sampling) to initiate the second MaaT033 treatment period of 28-day. At the end of the second Maat033 treatment period subjects will come to the study site (clinical examination, blood and feces sampling) and start a 28-day follow-up period without treatment.

Study completion is defined when all subjects enrolled completed the study follow-up period (clinical examination, blood and feces sampling) or earlier if a subject discontinued the study.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects aged between18 and 80 years
* ALS meeting the revised El Escorial criteria for possible, probable, laboratory-supported probable, or definite ALS (familial or sporadic)
* Time since first motor deficit at screening: at least 6 months, up to 24 months
* Slope of progression of ALS Functional Rating Scale - revised (ALSFRS-R) from date of symptom onset to date of screening test (ΔFS/number of months) between [0.4 and 1.1]
* Able to swallow study treatments (including capsules without opening or chewing them) as per the investigator's assessment
* SVC (Slow Vital Capacity) equal to or greater than 70% of the predicted normal value for sex, height, and age at the screening visit
* If taking riluzole, subject must be on a stable dose for ≥30 days
* Signature of written informed consent by subject

Exclusion Criteria:

* Subjects with a non-invasive ventilation, a tracheotomy and /or a gastrostomy
* Known autoimmune diseases, inflammatory disorders (SLE, Rheumatoid arthritis, connective tissue disorder) or chronic infections (HIV, hepatitis B, or C infection, Tuberculosis)
* Known hypersensitivity to rifaximin or macrogol or any of its components
* Known allergy or intolerance to trehalose, maltodextrin or Polyethylene Glycol (PEG)
* Documented hepatic impairment (Alanine Transaminase/ Aspartate Transaminase > 5N)
* Subject with white blood cells < 4000/ mm3; Polynuclear neutrophils < 1.5 G/ L
* Active infection requiring systemic antimicrobial therapy within 2-week prior to screening visit
* Active infection requiring systemic antimicrobial therapy between screening and baseline
* Medical condition requiring proton pump inhibitors (PPIs)
* Gastrointestinal obstruction or perforation
* Any gastro-intestinal bleeding in the past 3 months
* Gastric emptying disorders (gastroparesis)
* Toxic megacolon
* Severe forms of inflammation of the intestinal tract, including Crohn's disease and ulcerative colitis
* Severe vital organ dysfunctions unrelated to ALS and not compatible with experimental treatment, as per the investigator's assessment
* Subjects with negative IgG serology for Epstein Barr virus (EBV)
* Women of childbearing potential1 without effective contraceptive protection
* Nursing or pregnant women
* Any condition that, in the opinion of the investigator, may interfere with full participation in the study, including administration of study drug (and its preparation procedure) and attendance at required study visits; represent a significant risk to the subject; or interfere with the interpretation of study data
* Enrollment in another trial or expanded access program that may interfere with this study
* Guardianship/legal protection/curatorship of subjects
* Vulnerable subjects such as: persons deprived of liberty, persons in intensive care units unable to provide informed consent prior to the procedure

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2023-06-08 (Actual); Primary Completion 2024-07-22 (Actual); Study Completion 2024-07-22 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability: Incidence of Treatment Emergent Adverse Events (TEAE) grade >3, according to Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 | Day 84
  To assess the safety and tolerability of MaaT033 treatment

SECONDARY OUTCOMES:
Changes in gut microbiota profile | From Day -5 to Day 84 (at Day -5, Day 10, Day 28, Day 56 and Day 84)
  Analysis of fecal samples to assess gut microbiota alpha- and beta-diversity indices
Changes in levels of biomarkers in blood | From Day -5 to Day 84
  * Changes from baseline (Day -5) of neutrophil/ lymphocyte ratio, Interleukins (IL): IL-2, IL-6 and IL-8, Interferon gamma (IFNg), Tumor Necrosis Factor alpha (TNFa), Monocyte Chemoattractant Protein-1 (MCP-1), Transforming Growth Factor-beta (TGFb), the soluble subtype of CD14 (sCD14), C-reactive protein (CRP), erythrocyte sedimentation rate, plasma soluble Lipopolysaccharide Binding Protein (LBP), creatinin and serum Short-Chain Fatty Acids (SCFA) at Day 28, Day 56 and Day 84.
  * Changes from baseline (Day -5) of serum Neurofilament light (NfL) at Day 56 and Day 84.
Changes in levels of fecal calprotectin | From Day -5 to Day 84
  Changes from baseline (Day -5) of fecal calprotectin at Day 10, Day 28, Day 56 and Day 84

CONTACTS AND LOCATIONS:
Overall Officials: Gaelle Bruneteau, MD, PhD, Principal Investigator — Hôpital de la Pitié-Salpêtrière - CIC Neuroscience
Locations (2):
- France (2):
  - Centre Hospitalier Universitaire de Lille - CIC, Lille
  - Hôpital de la Pitié-Salpêtrière - CIC Neuroscience, Paris

IPD SHARING:
Plan to Share IPD: No